CLINICAL TRIAL: NCT00410449
Title: Study of the Effect of Oral Supplementation With Vitamin E on Circulating Oxidative Markers, Hemodialysis Vascular Access Occlusion, and Clinical Events in Patients With End Stage Renal Failure Treated by Hemodialysis
Brief Title: Oxidative Stress and Hemodialysis Access Failure
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Leonard B Rosenberg Renal Research Foundation (Unknown)
Other Study IDs: 11461-CP-001; NIEHS ES11461
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2006-12

CONDITIONS: End Stage Renal Disease; Hemodialysis
Keywords: End stage renal disease treated by hemodialysis; Hemodialysis vascular access patency; Vitamin E; oxidative markers; pentosidine; hydroxynonenal; levuglandin
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — alpha-Tocopherol

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Alpha tocopherol

SUMMARY:
Complications of hemodialysis access are the most frequent single reason for hospitalization among patients with End Stage Renal Disease (ESRD). Uremia, and particularly uremia in patients with diabetes, is a state of increased oxidative stress. The central hypothesis to be tested by this project is that oxidative stress is a major (and modifiable) trigger for vascular access complications. We hope to slow or reduce rates of stenosis, thrombosis and access complications by giving Vitamin E supplementation to patients being treated by hemodialysis.

DETAILED DESCRIPTION:
Patients continued their usual treatment on hemodialysis three times per week. This was a double-blinded placebo controlled trial. Patients took either Vitamin E 400 IU bid or placebo. An initial evaluation of access patency was performed and baseline blood drawn before starting Vitamin E. Every 3 months there was a followup evaluation with blood drawn for oxidative stress markers, and with a test of vascular access patency. The study was closed to new participants, vitamin E or placebo stopped, and data analysis performed in 2003.

ELIGIBILITY:
Inclusion Criteria:

Adults, end stage renal disease treated by hemodialysis, patent hemodialysis vascular access (graft or fistula)

Exclusion Criteria:

Temporary catheter dialysis access, inability to be compliant with study medication

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2001-05; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Miriam F Weiss, M.D., Principal Investigator — Case Western Reserve University
Locations (1):
- Center for Dialysis Care, Cleveland, Ohio, United States

REFERENCES:
- [Result] Schwing WD, Erhard P, Newman LN, Nodge MM, Czechanski BJ, Orlin SM, Walden SM, Behm K, Cacho CP, Negrea LA, Siu DS, Kern EO, Weiss MF. Assessing 24-hour blood glucose patterns in diabetic paitents treated by peritoneal dialysis. Adv Perit Dial. 2004;20:213-6. PMID 15384829